CLINICAL TRIAL: NCT02477410
Title: Effects of Hydrolysed Porcine Proteins on Muscle Protein Synthesis and Appetite
Acronym: SEPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Svineafgiftsfonden (Unknown); DC Ingredients (Unknown); Arla Food Ingredients Group P/S (Unknown)
Responsible Party: Principal Investigator, Arne Astrup, Prof., DM. DMSc., University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: H-15003581
Record Dates: First submitted 2015-06-11; First posted 2015-06-22 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Hunger; Satiety Response; Protein Synthesis
Keywords: porcine protein; appetite; muscle protein synthesis; gastrointestinal hormones

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hydrolysed porcine protein from blood (Experimental): Dietary intervention with hydrolysed porcine protein from blood
  Interventions: Dietary Supplement: Hydrolysed porcine protein from blood
- Hydrolysed porcine protein from muscle (Experimental): Dietary intervention with hydrolysed porcine protein from muscle
  Interventions: Dietary Supplement: Hydrolysed porcine protein from muscle
- Hydrolysed whey protein (Experimental): Dietary intervention with hydrolysed whey protein
  Interventions: Dietary Supplement: Hydrolysed whey protein

INTERVENTIONS:
Dietary Supplement: Hydrolysed porcine protein from blood — Effects of hydrolysed porcine proteins on muscle protein synthesis and appetite
  Arms: Hydrolysed porcine protein from blood
Dietary Supplement: Hydrolysed porcine protein from muscle — Effects of hydrolysed porcine proteins on muscle protein synthesis and appetite
  Arms: Hydrolysed porcine protein from muscle
Dietary Supplement: Hydrolysed whey protein — Effects of hydrolysed porcine proteins on muscle protein synthesis and appetite
  Arms: Hydrolysed whey protein

SUMMARY:
The purpose of the study is to obtain a better understanding of how hydrolysed porcine proteins affect the human metabolism, including the effects on muscle protein synthesis, appetite and secretion of gastrointestinal hormones.

It is hypothesised that hydrolysed porcine proteins will stimulate muscle protein synthesis, affect appetite and the secretion of gastrointestinal hormones similar to hydrolysed whey protein.

DETAILED DESCRIPTION:
Previous data show that proteins enhance satiety, decrease hunger and decrease energy intake. In addition, amino acids from dietary protein act as building blocks for de novo protein synthesis and consumption of dietary protein therefore stimulates protein synthesis. Proteins from different sources differ in amino acid composition and rate of absorption. Previously, studies on the effects of proteins on especially muscle protein synthesis has focused on milk proteins, whey and casein as animal sources, but other protein sources high in essential and branched-chain amino acids may also have beneficial effects on muscle protein synthesis and appetite. Thus, in this study the effects of two hydrolysed porcine proteins (one from porcine blood and one from porcine muscle) on muscle protein synthesis, appetite and secretion of gastrointestinal hormones will be compared with the effects of hydrolysed whey protein. These porcine proteins have never previously been tested and it is hypothesised that they may induce similar effects as hydrolysed whey protein due to the high contents of essential and branched-chain amino acids.

The study will be conducted as a randomised, 3-way, cross-over study. It consists of three visits separated by at least two weeks. It is expected that 18 normal-weight, young men will complete the study. They will be randomised to the order of the three proteins; hydrolysed porcine protein from blood (HPB), hydrolysed porcine protein from muscle (HPM) and hydrolysed whey protein (HW). At each visit the effects on muscle protein synthesis, appetite and secretion of gastrointestinal hormones will be measured/assessed. Muscle protein synthesis will be measured after consumption of a low (15 g) and a high (30 g) dose of protein and appetite and secretion of gastrointestinal hormones will be measured after the high protein dose (30 g). The effect on muscle protein synthesis will be measured by a flood-primed continuous infusion of labelled (Ring13C6) phenylalanine, muscle biopsies and blood samples. The effects on appetite will be assessed by visual analogue scales, an ad libitum meal and blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young men
* Normal weight (BMI 18.5-25 kg/m2)
* 22-40 years

Exclusion Criteria:

* Vegetarians
* Weight change >3kg within 2 months prior to start of the study
* Regular participation in cardio/strength training within 6 months prior to (and during) the study (>1 per wk)
* Use of alcohol >14 drinks/wk
* Drug abuse
* Smoking
* Regular consumption of protein supplements
* Use of over-the-counter or prescription medication that influences body weight, appetite or metabolism
* Diabetes Mellitus
* Dyslipidemia
* Diseases, which influence metabolism
* Donation of blood 3 months prior to start of (and during) the study
* Subjects with a hemoglobin value < 8 mol/L (measured at screening)
* Participation in other clinical studies 1 month prior to start of (and during) the study
* Subjects who are unable to give an informed consent.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in Muscle protein synthesis (%FSR) | 3 biopsies are taken at time 0, 150 min and 310 min at each visit
Change in Muscle protein synthesis (%FSR) | 13 blood samples are taken over 310 min

SECONDARY OUTCOMES:
Visual analogue scales (10 cm) | Assessed at time 0, 160, 175, 200, 220, 250, 280, 310, 345 min at each of the three test days
  Subjective appetite
Appetite - ad libitum energy intake | Measured once at time 325 min at each of the three test days
  At 325 min an ad libitum meal of spaghetti bolognese is served, and the total energy intake is recorded
Postprandial response in glycemic control, plasma amino acids and appetite regulating hormones | Blood samples are taken at 0, 150, 180, 200, 220, 250, 280 and 310 min at each of the three test days

OTHER OUTCOMES:
Urate in urine and blood | Blood samples are taken at 0, 20, 40, 60, 90, 120, 150, 180, 200, 220, 250, 280 and 310 min at each of the three test days. Urine is collected over 310 min at each test day
  Explorative parameter
Muscle protein breakdown, gene expression | 3 biopsies are taken at time 0, 150 min and 310 min. at each of the three test days
  Explorative parameter
Metabolomics - urine and blood | Blood samples are taken at 0, 20, 40, 60, 90, 120, 150, 180, 200, 220, 250, 280 and 310 min at each of the three test days. Urine is collected over 310 min at each test day
  Explorative parameter

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, DMSc, Principal Investigator — University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No